CLINICAL TRIAL: NCT03823066
Title: Experience With a Socially Assistive Robot for Home Care and Its Acceptance by People With Dementia, Caregivers and Dementia Trainers. A Mixed-method Intervention Study
Brief Title: Experience With a Robot for Home Care and Its Acceptance by People With Dementia, Caregivers and Dementia Trainers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Joanneum Research Forschungsgesellschaft mbH (Other); Sozialverein Deutschlandsberg (Unknown); Humanizing Technologies GmbH (Unknown)
Responsible Party: Principal Investigator, Sandra Schüssler, Deputy Head of the Institute of Nursing Science, Medical University of Graz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 30-401ex17/18a
Record Dates: First submitted 2019-01-09; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Dementia
Keywords: acceptance; usability; home care; socially assistive robot; humanoid robot; caregivers; dementia trainers; cognitive training; physical training
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: a humanoid socially assistive robot will be tested for people with dementia
Masking Description: not possible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coach Pepper (Experimental): Pepper is a humanoid socially assistive robot
  Interventions: Device: Coach Pepper

INTERVENTIONS:
Device: Coach Pepper — Robot Peppers's height is 1.20 meters and it weighs 28 kilograms. Pepper will be called Coach Pepper, because it is connected, via web interfaces, with a theratainment app including cognitive and physical training

SUMMARY:
Background:

Dementia rates are increasing worldwide and consequently burden global healthcare resources to a serious degree. However, there is a declining number of caregivers to provide care. It is for this reason that many new technologies, such as socially assistive robots, have been developed because of their potential to support caregivers in promoting the independence of people with dementia. Most of the (socially assistive) robots have so far been tested for people without dementia in mainly laboratory or institutional settings, like nursing homes. Consequently, there is a lack of knowledge about the possible uses of robots from the perspective of those affected by dementia in real-life/care situations (e.g. at home). Testing in a laboratory setting cannot capture the complexity and high variability of everyday situations occurring during the care of persons with dementia.

Methods

The design is a mixed method intervention study of a refined socially assistive humanoid robot. In total, three people with dementia, three relatives, three dementia trainers and three professional caregivers were included in the study. Quantitative data of technology acceptance were collected using the "Technology Usage Inventory". Qualitative data (main focus: experiences with the robot and handling the robot) were collected by means of observation and qualitative interviews. Movement data of people with dementia were collected by means of the eye camera of the robot.

This study helps to further refine and test a socially assistive robot for people with dementia living at home.

ELIGIBILITY:
Inclusion Criteria:

Persons with dementia:

* adults
* living at home
* all types of dementia
* light and moderate dementia (MMSE 10 and above)
* light dementia: living alone or with a relative at home (if alone: the relative should live in the neighborhood and be in daily contact with the person with dementia.)
* moderate dementia: living with a relative at home
* receive professional and/or non professional care or no care
* speak and understand German
* have no physical, auditory or visual restrictions, as this would make the application of the interventions impossible
* do not take any dementia-specific medication or have been taking dementia-specific medication for at least 3 months; condition stable and no change expected during the study period
* do not take antipsychotic and antidepressant medication or have been taking them for at least 14 days before study start
* children and pets in the household after previous individual discussion

Relatives:

* relatives of the participating persons with dementia (adults)
* relatives means family members, like spouse, daughter, aunt, ... or significant others like friends and neighbors
* living or not living with the person with dementia in the same household (in the case of moderate dementia, relatives must live in the same household)
* person with dementia receives or receives no professional care
* the relative provides or does not provide care
* If the person with dementia receives paid 24-hour care (regardless of whether they have mild or moderate dementia), a relative still has to be recruited as a participant (This relative must live in the same house or household and be in daily contact with the person with dementia).
* speak and understand German

Professional caregivers

* adults
* nurses
* speak and understand German

Dementia trainers

* adults
* trained as M.A.S. (Morbus Alzheimer Syndrome) trainer
* train the participants with dementia at home
* speak and understand German

ExclusioncCriteria:

Persons with dementia:

* known aggressive behavior
* frontotemporal Dementia

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2018-09-18 (Actual)

PRIMARY OUTCOMES:
Technology acceptance (all participants): "Technology Usage Inventory" | 1 week
  The questionnaire "Technology Usage Inventory" measures technology acceptance. It captures technology-specific and psychological factors contributing to the use of a technological device. The questionnaire has 8 dimensions (curiosity:4 items, anxiety:4 items, interest:4 items, usability/user-friendliness: 3 items, immersion:4 items, utility:4 items, skepticism:4 items and accessibility:3 items) with 30 items (7-point Likert scale). For every dimension 1- 21 or 28 points can be obtained. For all dimensions, higher levels on the respective dimension indicate a higher level of expression in the respective construct.
Experience with the robot (all participants) | 1 week
  Qualitative interviews with people with dementia. 1 qualitative focus group interview for all other participants.

SECONDARY OUTCOMES:
Handling the robot (people with dementia) | After 3 days of intervention
  Open, 1-hour semi-structured participant observation of people with dementia using the robot at home conducted by nurses.
Change of mobility (people with dementia) | 1 week
  Movement data collected by the eye camera of the robot.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Institute of Nursing Science, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] ADI. Journey of caring: an analysis of long-term care for dementia. ADI, London, 2013
- [Background] Bioethikkommission (Bioethics Commission). Roboter in der Betreuung alter Menschen - Stellungnahme der Bioethikkommission (Robots in the care of older people - statement of the Bioethics Commission). Geschäftsstelle der Bioethikkommission, Vienna, 2018
- [Background] Boman IL, Lundberg S, Starkhammar S, Nygard L. Exploring the usability of a videophone mock-up for persons with dementia and their significant others. BMC Geriatr. 2014 Apr 16;14:49. doi: 10.1186/1471-2318-14-49. PMID 24739662
- [Background] Lauriks S, Reinersmann A, Van der Roest HG, Meiland FJ, Davies RJ, Moelaert F, Mulvenna MD, Nugent CD, Droes RM. Review of ICT-based services for identified unmet needs in people with dementia. Ageing Res Rev. 2007 Oct;6(3):223-46. doi: 10.1016/j.arr.2007.07.002. Epub 2007 Aug 2. PMID 17869590
- [Background] Mao HF, Chang LH, Yao G, Chen WY, Huang WN. Indicators of perceived useful dementia care assistive technology: Caregivers' perspectives. Geriatr Gerontol Int. 2015 Aug;15(8):1049-57. doi: 10.1111/ggi.12398. Epub 2014 Nov 19. PMID 25407039
- [Background] NHI, WHO. Global Health and Aging http://www.who.int/ageing/publications/ global_health.pdf. Accessed 18. Dezember 2017, 2011.
- [Background] OECD. Adressing Dementia - the OECD response. OECD publishing, Paris, 2015.
- [Background] Pino M, Boulay M, Jouen F, Rigaud AS. "Are we ready for robots that care for us?" Attitudes and opinions of older adults toward socially assistive robots. Front Aging Neurosci. 2015 Jul 23;7:141. doi: 10.3389/fnagi.2015.00141. eCollection 2015. PMID 26257646
- [Background] Prince et al. World Alzheimer Report 2016 - Improving healthcare for people living with dementia. ADI, UK, 2016
- [Background] Robert Koch Institut. Gesundheit in Deutschland. Gesundheitsberichterstattung des Bundes (Health in Germany. Health report of the federal government). Gemeinsam getragen von RKI und Destatis. RKI, Berlin, 2015